CLINICAL TRIAL: NCT05424315
Title: Impact of DApagliflozin on Cardiac Function Following Anterior Myocardial Infarction in Non-Diabetic Patients - DACAMI (a Randomized Controlled Clinical Trial)
Brief Title: Impact of DApagliflozin on Cardiac Function Following Anterior Myocardial Infarction in Non-Diabetic Patients
Acronym: DACAMI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Omar Younis (Other Government)
Collaborators: Ain Shams University (Other)
Responsible Party: Sponsor-Investigator, Omar Younis, Clinical Research Coordinator, National Heart Institute, Egypt
Organization: National Heart Institute, Egypt (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTN1012021
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Anterior MI
Keywords: Heart Failure; Anterior MI; Dapagliflozin; Sodium Glucose Co-transporter 2 inhibitor; Anterior STEMI; Anterior ST Elevation Myocardial Infarction
MeSH Terms: conditions — Anterior Wall Myocardial Infarction; Heart Failure | interventions — dapagliflozin; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Active Comparator): Participants will receive Dapagliflozin 10mg once daily.
  Interventions: Drug: Dapagliflozin 10mg
- Control Group (Placebo Comparator): Participants will receive a glucose tab once daily.
  Interventions: Drug: Glucose Tab

INTERVENTIONS:
Drug: Dapagliflozin 10mg — 10mg Tab once daily
  Other Names: PubChem CID 9887712; BMS-512148; (1S)-1,5-anhydro-1-C-{4-chloro-3-[(4-ethoxyphenyl)methyl]phenyl}--glucitol; Forxiga; Edistride
  Arms: Intervention Group
Drug: Glucose Tab — Placebo Oral Tablet
  Other Names: PubChem CID 5793; D-Glucose; D-Glc
  Arms: Control Group

SUMMARY:
Sodium glucose co-transporter 2 inhibitors (SGLT2i) proved their favorable outcomes in heart failure. However, it is still unknown if their role extent into preventing heart failure, especially after acute myocardial infarction. This study aimed at identifying if there is such role for SGLT2i.

DETAILED DESCRIPTION:
A notable breakthrough in the management of heart failure is the use of a class of anti-diabetic medications known as, gliflozins. Gliflozins act by inhibiting the sodium glucose co-transporter 2 (SGLT-2). This is a transmembrane protein found at the luminal border of tubular cells of the proximal convoluted tubules of the kidney. It accounts for around 90% of glucose re-absorption. Inhibiting the SGLT-2 results in better glycemic control in patient with diabetes mellitus type 2 (DMT2).

In heart failure, sodium glucose co-transporter 2 inhibitors (SGLT2i - i.e., gliflozins) were found to have a favorable cardiovascular outcome independent of their anti-glycemic effect. In patients with acute myocardial infarction, the heart function as a pump is affected & heart failure develops. In particular, patients with anterior ST-elevation myocardial infarction (STEMI) are at a higher risk of remodeling & heart failure. This is due to the cutoff in blood supply in the left anterior descending (LAD) coronary artery which supplies a great area of left ventricle.

A question that rises: is there a role for SGLT2i, & in particular dapagliflozin, in acute myocardial infarction in improving post-infarction cardiac function & preventing heart failure? especially in patients who experience Anterior ST-Elevation Myocardial Infarction (STEMI).

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted with ECG Criteria for Anterior ST-elevation myocardial infarction according to the fourth universal definition of myocardial infarction*, ** & show echocardiographic evidence of reduced LV ejection fraction <50% & have undergone successful reperfusion by primary percutaneous coronary angiography (pPCI).

  * New ST segment elevation in contagious precordial leads consistent anatomically with the anterior wall of myocardium:

    * Men ≥ 40 years: 2 mV in leads V2-V3 &/or 1 mV in other precordial leads
    * Men <40 years: 2.5 mV in leads V2-V3 &/or 1 mV in other precordial leads
    * Women (regardless of age): 1.5 mV in leads V2-V3 &/or 1 mV in other precordial leads ** Patients with admission ECG showing DeWinter's Syndrome, Wellen Syndrome, New onset left bundle branch block, new onset right bundle branch block will also be included.

Exclusion Criteria:

1. Patients with Diabetes Miletus (Type 1 (DMT2), Type 1 (DMT1), secondary diabetes (e.g., endocrinopathies)
2. Patients already diagnosed with heart failure prior to this event
3. Patients on cardiotoxic chemotherapeutic medications.
4. Patients with haemoglobinopathies.
5. Patients with chronic organ damage (i.e., chronic hepatitis with MELD score >10, Stage 4 & 5 renal disease).
6. Patients already on SGLT2i.
7. Patients who will require additional anticoagulant therapy (i.e.: patients with transthoracic echocardiographic evidence of left ventricular thrombus).
8. Patients with contraindications for use of dapagliflozin including patients with severely impaired renal function (eGFR <30ml/min/1.73m2) &/OR previous history of genitourinary infections (i.e.: urosepsis, pyelonephritis & fournier's gangrene) &/OR at high risk of such infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
A change in NT-proBNP levels from baseline to 12 weeks post-anterior STEMI | 12 weeks
  Difference between both groups in the change of NT-proBNP levels from baseline to 12 weeks post-anterior STEMI
A change in left ventricular ejection fraction, end-diastolic volume or left ventricular mass index assessed by transthoracic echocardiography at baseline, 4 weeks & 12 weeks post-anterior STEMI | 12 weeks
  Difference between both groups in the change of the above mentioned echocardiographic parameters assessed at baseline, 4 weeks & 12 weeks post-anterior STEMI

CONTACTS AND LOCATIONS:
Overall Officials: Khairy Abdul-Dayem, M.D., Principal Investigator — Cardiology Department, Faculty of Medicine, Ain Shams University
Locations (2):
- Egypt (2):
  - Cardiology Department, Faculty of Medicine, Ain Shams University, Cairo
  - National Heart Institute, Cairo

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available through a data repository link provided to the publishing journal.
  Shared Data will include baseline characteristics of the intervention and control group. Moreover, NT-proBNP and Echocardiographic outcomes will be available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Access to the data will be feasible once the results are published.
Access Criteria: Access to the data will be feasible once the results are published after a formal request to the investigators. Approval of the the investigators is a must.

REFERENCES:
- [Result] Zinman B, Wanner C, Lachin JM, Fitchett D, Bluhmki E, Hantel S, Mattheus M, Devins T, Johansen OE, Woerle HJ, Broedl UC, Inzucchi SE; EMPA-REG OUTCOME Investigators. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2117-28. doi: 10.1056/NEJMoa1504720. Epub 2015 Sep 17. PMID 26378978
- [Result] Neal B, Perkovic V, Mahaffey KW, de Zeeuw D, Fulcher G, Erondu N, Shaw W, Law G, Desai M, Matthews DR; CANVAS Program Collaborative Group. Canagliflozin and Cardiovascular and Renal Events in Type 2 Diabetes. N Engl J Med. 2017 Aug 17;377(7):644-657. doi: 10.1056/NEJMoa1611925. Epub 2017 Jun 12. PMID 28605608
- [Result] Hummel CS, Lu C, Loo DD, Hirayama BA, Voss AA, Wright EM. Glucose transport by human renal Na+/D-glucose cotransporters SGLT1 and SGLT2. Am J Physiol Cell Physiol. 2011 Jan;300(1):C14-21. doi: 10.1152/ajpcell.00388.2010. Epub 2010 Oct 27. PMID 20980548
- [Result] Kalra S. Sodium Glucose Co-Transporter-2 (SGLT2) Inhibitors: A Review of Their Basic and Clinical Pharmacology. Diabetes Ther. 2014 Dec;5(2):355-66. doi: 10.1007/s13300-014-0089-4. Epub 2014 Nov 26. PMID 25424969
- [Result] McMurray JJV, Solomon SD, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Anand IS, Belohlavek J, Bohm M, Chiang CE, Chopra VK, de Boer RA, Desai AS, Diez M, Drozdz J, Dukat A, Ge J, Howlett JG, Katova T, Kitakaze M, Ljungman CEA, Merkely B, Nicolau JC, O'Meara E, Petrie MC, Vinh PN, Schou M, Tereshchenko S, Verma S, Held C, DeMets DL, Docherty KF, Jhund PS, Bengtsson O, Sjostrand M, Langkilde AM; DAPA-HF Trial Committees and Investigators. Dapagliflozin in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2019 Nov 21;381(21):1995-2008. doi: 10.1056/NEJMoa1911303. Epub 2019 Sep 19. PMID 31535829
- [Result] Packer M, Anker SD, Butler J, Filippatos G, Pocock SJ, Carson P, Januzzi J, Verma S, Tsutsui H, Brueckmann M, Jamal W, Kimura K, Schnee J, Zeller C, Cotton D, Bocchi E, Bohm M, Choi DJ, Chopra V, Chuquiure E, Giannetti N, Janssens S, Zhang J, Gonzalez Juanatey JR, Kaul S, Brunner-La Rocca HP, Merkely B, Nicholls SJ, Perrone S, Pina I, Ponikowski P, Sattar N, Senni M, Seronde MF, Spinar J, Squire I, Taddei S, Wanner C, Zannad F; EMPEROR-Reduced Trial Investigators. Cardiovascular and Renal Outcomes with Empagliflozin in Heart Failure. N Engl J Med. 2020 Oct 8;383(15):1413-1424. doi: 10.1056/NEJMoa2022190. Epub 2020 Aug 28. PMID 32865377
- [Result] Zannad F, Ferreira JP, Pocock SJ, Anker SD, Butler J, Filippatos G, Brueckmann M, Ofstad AP, Pfarr E, Jamal W, Packer M. SGLT2 inhibitors in patients with heart failure with reduced ejection fraction: a meta-analysis of the EMPEROR-Reduced and DAPA-HF trials. Lancet. 2020 Sep 19;396(10254):819-829. doi: 10.1016/S0140-6736(20)31824-9. Epub 2020 Aug 30. PMID 32877652
- [Result] Wright EM, Loo DD, Panayotova-Heiermann M, Hirayama BA, Turk E, Eskandari S, Lam JT. Structure and function of the Na+/glucose cotransporter. Acta Physiol Scand Suppl. 1998 Aug;643:257-64. PMID 9789568
- [Result] Shi L, Zhu D, Wang S, Jiang A, Li F. Dapagliflozin Attenuates Cardiac Remodeling in Mice Model of Cardiac Pressure Overload. Am J Hypertens. 2019 Apr 22;32(5):452-459. doi: 10.1093/ajh/hpz016. PMID 30689697
- [Result] Lee HC, Shiou YL, Jhuo SJ, Chang CY, Liu PL, Jhuang WJ, Dai ZK, Chen WY, Chen YF, Lee AS. The sodium-glucose co-transporter 2 inhibitor empagliflozin attenuates cardiac fibrosis and improves ventricular hemodynamics in hypertensive heart failure rats. Cardiovasc Diabetol. 2019 Apr 1;18(1):45. doi: 10.1186/s12933-019-0849-6. PMID 30935417
- [Result] Gaudron P, Eilles C, Kugler I, Ertl G. Progressive left ventricular dysfunction and remodeling after myocardial infarction. Potential mechanisms and early predictors. Circulation. 1993 Mar;87(3):755-63. doi: 10.1161/01.cir.87.3.755. PMID 8443896
- [Result] Santoro GM, Carrabba N, Migliorini A, Parodi G, Valenti R. Acute heart failure in patients with acute myocardial infarction treated with primary percutaneous coronary intervention. Eur J Heart Fail. 2008 Aug;10(8):780-5. doi: 10.1016/j.ejheart.2008.06.004. Epub 2008 Jul 2. PMID 18599344
- [Result] Masci PG, Ganame J, Francone M, Desmet W, Lorenzoni V, Iacucci I, Barison A, Carbone I, Lombardi M, Agati L, Janssens S, Bogaert J. Relationship between location and size of myocardial infarction and their reciprocal influences on post-infarction left ventricular remodelling. Eur Heart J. 2011 Jul;32(13):1640-8. doi: 10.1093/eurheartj/ehr064. Epub 2011 Mar 12. PMID 21398642
- [Derived] Dayem KA, Younis O, Zarif B, Attia S, AbdelSalam A. Impact of dapagliflozin on cardiac function following anterior myocardial infarction in non-diabetic patients - DACAMI (a randomized controlled clinical trial). Int J Cardiol. 2023 May 15;379:9-14. doi: 10.1016/j.ijcard.2023.03.002. Epub 2023 Mar 6. PMID 36889650